CLINICAL TRIAL: NCT04375345
Title: A Retrospective Study Evaluating Clinical and Radiographic Early Outcomes of Total Hip Arthroplasty and Revision Hip Arthroplasty With DELTA Multihole TT Cup.
Brief Title: DELTA Multihole TT Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Bratislava (Other)
Responsible Party: Principal Investigator, Boris Steno, Boris Steno MD PhD Assoc Prof, University Hospital Bratislava
Other Study IDs: UHBratislava
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Hip Osteoarthritis; Arthroplasty Complications; Hip Dysplasia
Keywords: total hip arthroplasty; hip arthroplasty revision; complex primary arthroplasty; trabecular titanium
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Dislocation | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: hip arthroplasty — complex primary total hip arthroplasty or revision total hip arthroplasty performed through anterolateral or posterolateral approach
  Other Names: revision hip arthroplasty

SUMMARY:
A retrospective study evaluating clinical and radiographic early outcomes of total hip arthroplasty and revision hip arthroplasty with DELTA Multihole TT cup.

ELIGIBILITY:
IInclusion criteria as per DELTA Multihole TT indications for use:

Age ≥ 18 years

* Non-inflammatory degenerative joint disease such as osteoarthritis or avascular necrosis;
* Signed Informed consent
* Hip dislocation using protruded liners, spacers;
* Rheumatoid arthritis;
* Post-traumatic arthritis;
* Correction of functional deformity in case of acetabulum verticalization, anteversion, and retroversion;
* Fractures of femoral neck;

If used in combination with spacers and hemispheric modules, other indications are:

* Revision of previous unsuccessful femoral head replacement, cup arthroplasty or other procedure;
* Clinical management problem where arthrodesis or alternative reconstruction techniques are less likely to achieve satisfactory results;
* Where bone stock is of poor quality or is inadequate for other reconstruction techniques as indicated by deficiencies of the acetabulum.

Exclusion criteria as per DELTA Multihole TT contraindications for use:

* Local or systemic infections;
* Septicaemia;
* Persistent acute or chronic osteomyelitis;
* Confirmed nerve or muscle lesion compromising hip joint function;
* Vascular or nerve diseases affecting the concerned limb;
* Poor bone stock compromising the stability of the implant;
* Metabolic disorders which may impair fixation and stability of the implant;
* Any concomitant disease and dependence that might affect the implanted prosthesis;
* Metal hypersensitivity to implant materials.

Additional exclusion criteria:

• Female patients who are pregnant, nursing, or planning a pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from patients who underwent a Total Hip Arthroplasty with the DELTA Multihole TT cup. Both complex primary and revision cases are considered.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-23 (Actual); Primary Completion 2022-01-23 (Estimated); Study Completion 2022-03-23 (Estimated)

PRIMARY OUTCOMES:
Percentage of HHS score equal or greater than "Good" at 2 years after surgery | Month 24

SECONDARY OUTCOMES:
Radiographic implant evaluation and stability assessment | Week 6, Week 12, Month 6, Month 12, Month 24
  Migration over 2 mm or over 5 degrees
Survival rate | Month 24
  Kaplan-Meier
Patients recovery at 2 years after surgery evaluated using the 5-level EQ-5D version (EQ-5D-5L). | Month 24
  The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
Incidence of device-related Adverse Events / Serious Adverse Events | Intraoperative, Week 6, Week 12, Month 6, Month 12, Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Boris Steno, MD PhD Prof, Principal Investigator — University Hospital Bratislava
Locations (1):
- 2nd University Department of Orthopaedic and Trauma Surgery Comenius University Faculty of Medicine, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No